CLINICAL TRIAL: NCT04152343
Title: An Intraoperative Guidance Platform for Radio Frequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Eric K. Hoffer, Director, Vascular and Interventional Radiology, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SF19108; 2R44CA189515 (NIH)
Record Dates: First submitted 2019-11-02; First posted 2019-11-05 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Radiofrequency Ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- RFA Physics Library- PGP (Experimental): The RFA Physics Library will be used during during percutaneous liver RFA procedures.
  Interventions: Device: RFA Physics Library -- a Planning and Guidance Platform (PGP)

INTERVENTIONS:
Device: RFA Physics Library -- a Planning and Guidance Platform (PGP) — Research software used to support liver RFA of HCC lesions >2cm

SUMMARY:
This study tests the hypothesis that use of the research RFA (Radiofrequency ablation) Physics Library will result in more frequent technical success (complete necrotization of target tissues) compared to ablations conducted without computer guidance.

The RFA Physics Library -- a Planning and Guidance Platform (PGP) (NE Scientific, LLC) -- will be used to support percutaneous liver RFA under CT-guidance by assisting physicians in the identification of ablation targets, assessment of proper ablation probe placement, and projection of the created ablation zones on the CT image.

DETAILED DESCRIPTION:
Patients referred for curative ablation of an HCC by consensus recommendation of the multidisciplinary Liver Tumor Clinic at a 400-bed academic cancer center from June 2018 through December 2021 were considered for participation in the study.

Inclusion criteria :

patient : over 18 years old , ble to provide informed consent, expected survival >1 year lesion: HCC, >2 cm in diameter, located > 1 cm from any other lesion. procedure : completed using the support of the Accublate simulation software.

Software detail at : Hoffer EK, Borsic A, Patel SD. Validation of Software for Patient-Specific Real-Time Simulation of Hepatic Radiofrequency Ablation. Acad Radiol. 2022 Oct;29(10):e219-e227. doi: 10.1016/j.acra.2021.12.018. PMID: 35039220; PMCID: PMC9276838

Treatment: CT-guided RFA with Boston Scientific LeVeen system, RF3000 Generator. .

Prophylactic antibiotic General anesthesia; imaging during suspended ventilation, no PEEP Ablation per manufacturer's protocol. Target : tumor + 5 mm margin Planning, targeting, intraprocedural repositioning, assessment of ablation coverage using software simulation in conjunction with manufacturer's data map.

Tract ablation

Follow-up clinic visit with contrast-enhanced cross-sectional imaging (MRI or CT) at 3 months, then every 3 months x 2 years. Data review for complications, progression of liver disease, evidence of local, regional, or metastatic disease, and additional interventions.

Outcome measures: primary : local tumor progression secondary: hepatic tumor progression

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Presence of hepatocellular carcinoma with a size equal or larger than 2cm.
3. Scheduled for CT-guided thermal ablation under General Anesthesia
4. Able to provide written, informed consent

Exclusion Criteria:

1. Absolute of relative contraindication to MRI:

   1. the presence of an electronic implant, such as a pacemaker not approved for MRI
   2. the presence of a metal implant, such as an aneurysm clip not approved for MRI
   3. claustrophobia
   4. the presence of other contraindication(s), such as inability to comfortably lie flat, history of working with metal, other implanted hardware or shrapnel
2. Target tumor adjacent to or within prior ablated or resected site.
3. Serious psychiatric illness not adequately controlled to permit patient cooperation to obtain an MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-12-07 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric K Hoffer, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients referred from multidisciplinary Liver Tumor Clinic from 12/2019-12/2021 with a lesion consistent with HCC (AASLD criteria) > 2 cm diameter, were offered participation in study
Pre-assignment Details: Five enrolled were excluded: 4 based on pre-procedure study demonstrating tumor outside criteria (2 < 2 cm, 2 > 6 cm diameter); one patient excluded due to technical factors precluding connection of software.
Units Other Than Participants: tumors
Groups:
- RFA Physics Library- Ablation Simulation Guidance: The RFA Physics Library -- a Planning and Guidance Platform: Research software will be used during percutaneous liver RFA of HCC lesions >2cm
Period: Overall Study
Arm/Group | RFA Physics Library- Ablation Simulation Guidance
Started | 57; 68 tumors (57 procedures in 52 unique patients (patients could be re-enrolled for new tumor at least 2 cm from prior treated lesion))
Completed Procedure | 57; 68 tumors
Completed 2-3 m Imaging for Efficacy | 57; 68 tumors (assessment of complete ablation : no evidence for residual enhancement of tumor or within 1 cm on CT or MRI.)
Completed (completed 2 year enhanced MRI/CT follow-up) | 29; 37 tumors
Not Completed | 28; 31 tumors
Not completed — Transplanted | 5
Not completed — Death | 20
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: patients/tumors that were treated using ablation simulation guidance software
Units Other Than Participants: tumors
Groups:
- Patients: patients enrolled and had HCC treated with RFA utilizing Ablation Simulation Guidance software
Arm/Group | Patients
Number analyzed (Participants) | 57
Number analyzed (tumors) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 55
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 57
Cirrhosis Etiology [Number; unit: participants]
  Hepatitis C | 28
  Hepatitis B | 3
  Alcohol | 36
  Metabolic dysfunction-associated steatohepatitis | 19
  other | 2
Child Turcotte Pugh Class [Count of Participants; unit: Participants] — Child-Turcotte-Pugh score correlates with operative risk for cirrhotic patients. It is calculated from clinical signs/findings:
  Ascites : none: 1, diuretic responsive: 2, diuretic refractory: 3 Hepatic encephalopathy : none: 1, controlled with medications: 2, not controlled; 3 total bilirubin (mg/dl). <2 : 1, 2-3 : 2, >3 : 3 albumin (g/dl): >3.5 : 1, 2.8-3.5 : 2, < 2.8 : 3 international normalized ratio: < 1.7: 1, 1.7-2.3 : 2, >2.3 : 3
  The higher total points correlate with increased mortality risk:
  5-6 points : class A 7-9 : B 10-15. : C
  Participants
    A | 32
    B | 18
    C | 7
Functional Status (ECOG) [Count of Participants; unit: Participants] — Performance Status was evaluated by the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale:
  0: fully active
  1. no strenuous
  2. activities of daily living (ASL), no work, up>50% of day
  3. limited ADL, in chair > 50% of day
  4. no ADL, confined to bed/chair
  5. dead
  Participants
    0 | 39
    1 | 16
    2 | 2
Tumor burden per patient [Number; unit: participants] — count of tumors treated in each participants treatment session
  participants
    1 tumor | 43
    2 tumors | 8
    3 tumors | 4
    5 tumors | 2
Alpha Fetoprotein > 20 ng/ml [Count of Participants; unit: Participants] — alpha fetoprotein (AFP) above institutional normal limit.
  Participants | 8
Prior Hepatocellular Carcinoma treatment [Count of Participants; unit: Participants] — number of patients previously treated for HCC by ablation, surgery, chemotherapy or radiation therapy
  Participants | 36
Within MIlan criteria [Count of Participants; unit: Participants] — Milan criteria are that the hepatocellular carcinoma is limited to 3 tumors < 3 cm in diameter or a single tumor < 5 cm in diameter, without evidence for lymphadenopathy, metastasis or vascular involvement. Beyond these limits, the HCC is considered unacceptable for liver transplant due to risk of recurrence.
  Participants | 46
Tumor Size [Mean (Inter-Quartile Range); unit: centimeters] | 2.73 [2.2 to 3.1]
Biopsy Grade [Count of Participants; unit: Participants] — histopathologic grade based on World Health Organization classification. Gisder DM, Tannapfel A, Tischoff I. Histopathology of hepatocellular carcinoma - when and what. Hepatoma Res 2022;8:4. http://dx.doi.org/10.20517/2394-5079.2021.106
  Participants
    well-differentiated | 16
    moderately-differentiated | 17
    poorly-differentiated | 5
    not available (LIRADS 5) | 19
Liver segment location [Count of Units; unit: tumors]
  segment II | 3
  segment III | 13
  segment IV | 7
  segment V | 9
  segment VI | 8
  segment VII | 12
  segment VIII | 16

OUTCOME MEASURES:

1. Primary Outcome: Rate of Technical Success of Tumor Ablation
Description: Technical success is defined as the complete ablation of the target lesion (tumor and 5 mm margin), as determined by operator.
Time Frame: Success measured at end of RFA procedure, one-time event (lasting up to a few hours)
Population: tumors completely treated (tumor + >95% of 5 mm margin)
Measure: Count of Units; unit: tumors
Units Other Than Participants: tumors
Groups:
- Tumors Treated With Ablation Simulation Guidance.: The RFA Physics Library -- a Planning and Guidance Platform: Research software will be used during percutaneous liver RFA of HCC lesions >2cm
Arm/Group | Tumors Treated With Ablation Simulation Guidance.
Number analyzed (Participants) | 57
Number analyzed (tumors) | 68
tumors
  complete | 68
  incomplete | 0

2. Primary Outcome: Rate of Local Tumor Recurrence
Description: Local recurrence at 2 years is defined as the detection of viable malignant tissues at edge of or within a site which was previously treated by RFA.
Time Frame: 2 years after RFA treatment
Population: KM evaluation for proportion with local recurrence at 2-year follow-up
Measure: Count of Units; unit: tumors
Units Other Than Participants: tumors
Arm/Group | Tumors Treated With Ablation Simulation Guidance.
Number analyzed (Participants) | 57
Number analyzed (tumors) | 68
tumors
  local recurrence at 2 years | 9
  no local recurrence at 2 years | 59

ADVERSE EVENTS:
Time Frame: within 30 days of procedure
Description: Adverse events were evaluated based on whether suspected/potentially related to the use of guidance software for the ablation versus the ablation procedure versus underlying patient disease/comorbidities.
  Adverse event collection based on patient clinical follow up during first month and then at 3 month clinic visits.
Groups:
- Ablation Simulation Guidance: The RFA Physics Library -- a Planning and Guidance Platform software was used to provide ablation simulation guidance to support liver RFA of HCC lesions >2cm
Arm/Group | Ablation Simulation Guidance
All-Cause Mortality (participants affected / at risk) | 20/57
Serious Adverse Events (participants affected / at risk) | 2/57
Other Adverse Events (participants affected / at risk) | 4/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablation Simulation Guidance (N=57)
hypotension (Injury, poisoning and procedural complications) | 1 (1) — hypotension with altered mental status in recovery and CT identified a large subcapsular hematoma at the subcapsular ablation site that requried ICU and 2 unit transfusion; definitely procedural related, unclear relation to software use
hypoglycemia (Nervous system disorders) | 1 (1) — re-admission 3 days after ablation for mental status changes due to difficult-to-control hypoglycemia. Probably medication-related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablation Simulation Guidance (N=57)
mild-moderate : urinary retention (Renal and urinary disorders) | 4 (4) — urinary retention in 3 males, 1 female. Required additional day stay (n=2) discharge with Foley catheter, Urology follow-up. Related to ablation procedure but not use of software guidance.

LIMITATIONS AND CAVEATS:
Limited by no comparative cohort, small numbers (high drop out due to mortality before 2 yrs).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT04152343/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT04152343/SAP_001.pdf